CLINICAL TRIAL: NCT04270123
Title: An International Phase 4 Field Study to Analyse the Psychometric Properties of the Updated Module on Assessing Quality of Life of Patients With Breast Cancer (EORTC QLQ-BR23, Update EORTC QLQ-BR45)
Brief Title: An EORTC Study Updating the QLQ-BR23 to BR45
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Principal Investigator, Galina Velikova, Professor of Psycho-social and Medical Oncology/Consultant in Medical Oncology, University of Leeds
Other Study IDs: 275142
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Cancer; Breast Cancer
Keywords: EORTC; PRO; PROM; Adverse Event; Quality of Life
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 consists of breast cancer patients with local or locally advanced disease. All participants will complete the EORTC QLQ-C30 and BR-45 questionnaires. A subgroup of participants within this group (those who have changed disease or treatment status) will be asked to complete the above questionnaires again, three months later (+-1 week). They will also complete an anchor question. Completing twice is for the responsiveness to change analysis.
  Interventions: Other: EORTC QLQ-BR45 questionnaire
- Group 2: Group 2 consists of metastatic breast cancer patients. All participants will complete the EORTC QLQ-C30 and BR-45 questionnaires at one time point only.
  Interventions: Other: EORTC QLQ-BR45 questionnaire
- Group 3 - follow up: Group 3 consists of follow up breast cancer patients. All participants will complete the EORTC QLQ-C30 and BR-45 questionnaires. One-to two weeks later, a subgroup of participants in this group (with no evidence of disease and /or change in health status) will complete the above questionnaires, as well as an anchor question. Completing twice is for the test-retest analysis.
  Interventions: Other: EORTC QLQ-BR45 questionnaire

INTERVENTIONS:
Other: EORTC QLQ-BR45 questionnaire — The EORTC QLQ-BR23 questionnaire has been updated with a further twenty-two items to create the EORTC QLQ-BR45. This updated questionnaire contains items to encapsulate advancements in knowledge about the epidemiology of breast cancer and side effects experienced with new treatments. This study will test the psychometric properties of the EORTC QLQ-BR45 as a measure of quality of life in patients with breast cancer.

SUMMARY:
Female breast cancer is still the most frequent type of cancer in Europe with 21 per 100,000 women .The EORTC QLQ-BR23 was one of the first modules developed to be used in conjunction with the core questionnaire EORTC QLQ-C30 and was published in 1996. Since the beginning of the work on the EORTC QLQ-BR23 some 20 years ago, much knowledge has been gathered about the epidemiology of breast cancer, and major advances have been made with regard to diagnostic and therapeutic options. Therefore, the EORTC Quality of life group decided to update the BC23. A phase 1 to 3 module development project has been completed. This resulted in a 45 item module, retaining 23 of the original items and adding 22 new items, particularly tapping into the side effects of new systemic and local therapies.

The aim of the Phase 4 study is to test the scale structure, reliability, responsiveness to change, and validity of the EORTC QLQ-BC45 in conjunction with the EORTC QLQ-C30 in patients diagnosed with breast cancer. Participants will be enrolled in four groups according to their disease stage (1. local/locally advanced disease, 2. metastatic disease, 3. follow up. Various combinations of therapies are permissible.

According to sample size calculations, we will include a total of N =490 patients from 12 countries.

Participants will be invited to complete the QLQ-C30 and the QLQ-BC45, followed by the Debriefing Questionnaire. Data of all patients will be used to evaluate the scale structure, internal consistency, convergent and discriminant validity. A subgroup of follow up patients with no evidence of disease (no change in health status) will be invited to complete the QLQ-C30 and the QLQ-BC45 for a second time one to two weeks later for the test-retest analysis. A subgroup of patients from the local/ locally advanced breast cancer group (who have had change in disease or treatment status after the first assessment) will be invited to complete a second set of questionnaires for the response to change analysis. Sociodemographic and clinical data will be recorded using standardized case report forms (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Adult females aged 18 years or over
* Histologically confirmed diagnosis of breast cancer (any type) with no previous primary or recurrent tumour
* Receiving or have previously received curative or palliative treatment.
* Able to understand/speak English and complete the questionaires
* Have the capacity/mental fitness to give written informed consent and complete the questionnaires.

Exclusion Criteria:

* Male gender or transgender
* Inability to understand/speak English and complete the questionnaire
* Patients with any psychiatric condition or cognitive impairment, as determined by the treating physician, that would hamper participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
EORTC-BR45 questionnaire | 2020-2021
  This is a questionnaire validation study. No reporting score on scale.

CONTACTS AND LOCATIONS:
Overall Officials: Galina Velikova, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Webpage with brief study description — https://qol.eortc.org/questionnaire/update-qlq-br23/